CLINICAL TRIAL: NCT00442351
Title: A Comparative Study of The Efficacy and Tolerability of Maintenance Treatment of Patients With Mild/Moderate Persistent Asthma With Asmanex Twisthaler 220 mcg QD PM Versus "Asmanex" Placebo QD PM
Brief Title: Efficacy and Tolerability of Maintenance Treatment With Asmanex Twisthaler Versus Placebo in Mild/Moderate Persistent Asthmatics (Study P04654)(TERMINATED)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow Enrollment
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04654; IND Number: 46216; SCH 032088 (Registry Identifier: NCT00442351)
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Results first posted 2010-04-16 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asmanex Twisthaler (Experimental)
  Interventions: Drug: Asmanex twisthaler
- Placebo inhaler (Placebo Comparator)
  Interventions: Other: Placebo for Asmanex twisthaler

INTERVENTIONS:
Drug: Asmanex twisthaler — Asmanex Twisthaler 220 mcg provided once daily in the evening for 12 weeks
  Other Names: Mometasone furoate inhalation powder
  Arms: Asmanex Twisthaler
Other: Placebo for Asmanex twisthaler — Placebo for Asmanex Twisthaler 220 mcg, once daily in the evening for 12 weeks
  Arms: Placebo inhaler

SUMMARY:
This is a randomized, multicenter, placebo-controlled, double-blind, parallel-group study evaluating Asmanex Twisthaler 220 mcg once daily (QD) in the evening (PM) compared with "Asmanex" Placebo QD PM for 12 weeks. Efficacy will be measured for the changes in forced expiratory volume in 1 second (FEV1) from baseline to the end of treatment period (Week 12 or end of the study).

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent
* Be 18-75 years of age, of either sex and any race
* Have asthma for >= 12 months
* Have mild or moderate persistent asthma
* Prior to completing Screening Visit procedures, must be using: low or moderate doses of an inhaled corticosteroid (IC), with a short-acting beta-2 agonist (SABA) as needed (prn) or a SABA prn as monotherapy. Those using a combination ICs plus long-acting beta-2 agonist (LABA) medication, such as Advair 100/50 twice daily (BID), must be changed to fluticasone propionate 100 mcg BID for at least 5 days prior to the start of Run-In-Period. Those using LABA as monotherapy must be switched to SABA prn for at least 5 days prior to the start of Run-In Period
* Be off treatment with leukotriene receptor antagonist (LTRA) for at least 14 days prior to Screening
* Have an FEV1 >=65% but <=85% of predicted normal value at Screening and at Baseline when SABAs have been withheld for at least 6 hours
* Demonstrate an increase of absolute FEV1 of >= 12% with an absolute volume increase of at least 200mL during Screening. Written documentation of FEV1 reversibility of >= 12% within 2 years prior to Screening was acceptable in lieu of testing. FEV1 reversibility testing should be done after withholding inhaled SABA for at least 6 hours
* Have a frequency of asthma score of at least 2 (at least 2 symptoms) and/or frequency of bronchodilator use score of at least 2 at Screening
* Have a Total Asthma Severity Score (TASS) of at least 4 on 8 or more of the AM and PM recordings from the last 7 days during the Run-in period prior to Baseline and the AM of the Baseline Visit
* At Screening Visit, have sleep disturbance and scores of >=2 on the interference with sleep rating scale (recall over the past 7 nights), and at least 30 on the Medical Outcomes Study Sleep scale (MOS-SS) Sleep Disturbance Sleep Scale (recall over the past 7 days)
* At the Baseline Visit, must have sleep disturbance and scores of >= 2 on interference with sleep rating scale (recorded in a diary during the past 7 nights), and at least 30 on the MOS-SS Sleep Problems Index II 9 items(SLP 9)

Exclusion Criteria

* Women who are pregnant or intend to become pregnant during the study
* Women who are nursing or intend to nurse during the study or within 30 days after completion
* Have participated in any clinical trial within the last 30 days or in one involving antibodies for asthma or rhinitis within 3 months prior to Screening
* Have had an unscheduled medical visit (due to exacerbation of asthma) within 1 month prior to Screening
* Have been treated in the emergency room or admitted to the hospital due to exacerbation of asthma on two or more occasions within the 12 months prior to Screening
* Have used >12 puffs of rescue SABAs or 2 treatments with a nebulized beta-2-agonist per day on 2 consecutive days within 4 weeks prior to Screening
* Required more than 2 courses of oral/systemic corticosteroids for asthma within 12 months prior to Screening
* Have a history of sleep disorders, including narcolepsy, or use of medications that affect alertness or sleep
* Have sleep apnea, obstructive sleep apnea-hypopnea, or are being treated with the ventilation devices Continuous Positive Airway Pressure (CPAP) or (Bi-level Positive Airway Pressure (Bi-PAP), or are receiving oxygen by inhalation
* Are smokers or ex-smokers who have smoked within 6 months prior to

Screening or have a cumulative smoking history of 10 pack-years or greater

* Are allergic to corticosteroids, SABAs, or LABAs
* Required ventilator support for respiratory failure secondary to asthma in the last 10 years
* Have a Body-Mass-Index greater than 35

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Inhaler: Placebo for Asmanex Twisthaler 220 mcg, provided once daily in the evening for 12 weeks
Period: Overall Study
Arm/Group | Asmanex Twisthaler | Placebo Inhaler
Started | 17 (Due to poor enrollment and a high screening failure rate, this study was terminated early.) | 9
Completed | 10 | 3
Not Completed | 7 | 6
Not completed — Administrative | 6 | 5
Not completed — Did not meet protocol eligibility | 1 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asmanex Twisthaler | Placebo Inhaler | Total
Number analyzed (Participants) | 17 | 9 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 8 | 25
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (11.9) | 42.6 (17.0) | 42.1 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 7 | 2 | 9
Region of Enrollment [Number; unit: participants]
  United States | 17 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Final/Terminal Visit in Forced Expiratory Value in 1 Second (FEV1) in Morning Office Measurements.
Description: The baseline value for this outcome measure was evaluated at the baseline visit prior to randomization. The change from Baseline to final/terminal visit in FEV1 was to be analyzed using an Analysis of Covariance (ANCOVA) model.
Time Frame: Twelve (12) weeks
Arm/Group | Asmanex Twisthaler | Placebo Inhaler
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Asmanex Twisthaler | Placebo Inhaler
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/9
Other Adverse Events (participants affected / at risk) | 5/17 | 3/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Asmanex Twisthaler (N=17) | Placebo Inhaler (N=9)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Scar excision (Surgical and medical procedures) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was terminated early due to a high screening failure rate and poor enrollment that resulted from stringent inclusion and exclusion criteria. Efficacy data were not evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is not allowed to release any interim results of the Study without prior consent of the sponsor, and must provide 45 days written notice to the sponsor prior to public release to permit the sponsor's review. The PI can use the study results for his/her own teaching, research, and publication purposes only, not for commercial purposes, except as authorized by the sponsor. No publication shall contain any trade secret or proprietary/confidential information of the sponsor.